CLINICAL TRIAL: NCT04294381
Title: Achievement and Adherence to Behavioral Health Goals in the Setting of Patient-Directed Goal Choice
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Donna R Zwas, Senior Cardiologist, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HMO0094-15
Record Dates: First submitted 2019-10-27; First posted 2020-03-04 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Sedentary Behavior; Risk Reduction
MeSH Terms: conditions — Sedentary Behavior; Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: evaluation of tablet-based decision tool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pilot of SMART-goal-setting health behavior decision tool (Experimental): participants will be asked to use a decision tool to choose and delineate SMART health behavior goals
  Interventions: Behavioral: Decision tool

INTERVENTIONS:
Behavioral: Decision tool — participants will be asked to use a decision tool to choose and delineate SMART health behavior goals

SUMMARY:
Health care decisions should include patients' health outcome goals and care preferences so as to enable a unified set of individualized patient outcome goals, rather than disparate disease-specific goals that do not reflect patient choice and commitment. This study utilizes a skilled professional interview and a simple tablet-based tool to enable patient choice of health behavior goals. The tool guides the patient to choose a specific, measurable, attainable, realistic and time-based (SMART) goal. The hypothesis of this study is that the implementation this patient choice tool will increase the likelihood of patient adherence to the goal and increase patient self efficacy.

DETAILED DESCRIPTION:
Health care decisions should include patients' health outcome goals and care preferences so as to enable a unified set of individualized patient outcome goals, rather than disparate disease-specific goals that do not reflect patient choice and commitment. This study utilizes a skilled professional interview and a simple tablet-based tool to enable patient choice of health behavior goals. The tool guides the patient to choose a specific, measurable, attainable, realistic and time-based (SMART) goal. The hypothesis of this study is that the implementation this patient choice tool will increase the likelihood of patient adherence to the goal and increase patient self efficacy.

Patients who participate in the Women's Heart Clinic at Hadassah will be recruited to participate in the study. Patients are to be included in this study if they have undergone cardiovascular event (myocardial infarction, percutaneous coronary intervention, or stroke,) had an active cardiac symptom (e.g. chest pain or arrhythmia) or had three or more active risk factors (i.e. diabetes, hypertension, hyperlipidemia, peripheral artery disease, current smoker, family history of premature coronary disease, gestational diabetes, pregnancy-induced hypertension/pre-eclampsia, or obesity). Patients are excluded if they arere pregnant, have type 1 diabetes, a psychiatric diagnosis that precluded participation, dementia, or if they were under the care of another multi-disciplinary clinic. The Hadassah Heart Center for Women follows a team-based approach, consisting of a cardiologist, nurse/coordinator, nutritionist, physical therapist/exercise expert and psychologist. At the first visit, patients met with all five professionals. The nurse/coordinator interviews the patient and assists in baseline data collection. The physician obtains the history, conducted physical examinations and determined cardiac care plans. The nutritionist assesses the patient's diet and assists the patient with determining SMART (specific, measurable, achievable, realistic and time-bound) goals using the table tool. The physical therapist/exercise expret performs an assessment of physical activity capacity and behaviors,a 6 minute walk test, and assists the patient in determining SMART goals for increased physical activity. The psychologist assessed patient for active mental health concerns that would interfere with self-care, assisted her in developing a plan to maximize self-care and developed a referral plan for patients who required mental health intervention. Patient cases are reviewed in a multi-disciplinary meeting after the visit and a comprehensive letter including specific recommendations from each member of the team was sent to the patient (In Israel, letters are given to the patient rather than directly to the referring physician.) Follow up appointments are scheduled according to clinical indications.

Baseline data collection included age, medical history, country of birth, education, and monthly income. Cardiac risk factors included the inclusion criteria as described above.

Health behaviors including nutrition behaviors, physical activity behaviors, smoking and alcohol consumption are measured using a culturally-adapted translation of the Healthy Heart Score and Mediterranean Diet Score. The patients fill out the Depression, Anxiety, Stress Score and the Brief Experiential Avoidance Score, health self efficacy and overall quality of life.

Patients will be followed by telephone/video conference at 1 and 2 months, return for follow up visit at month 3, telephone/video conferecnce follow up will be done at months 4 and 5, and the patient will return at month 6 for outcomes evaluation, which will include nutrition and physical activity assessment, and health self efficacy, Health Heart Score, Brief Experiential Avoidance Score, and Health self efficacy. In case of corona restrictions, visits 3 and 6 may be done remotely as well

ELIGIBILITY:
Inclusion Criteria:

* females age 18-90
* who fall into one of the following categories:

  * undergone cardiovascular event (myocardial infarction, percutaneous coronary intervention, or stroke,) or
  * who have an active cardiac symptom (e.g. chest pain or arrhythmia) or
  * have three or more active risk factors (i.e. diabetes, hypertension, hyperlipidemia, peripheral artery disease, current smoker, family history of premature coronary disease, gestational diabetes, pregnancy-induced hypertension/pre-eclampsia, or obesity).

Exclusion Criteria:

* pregnancy
* type 1 diabetes
* a psychiatric diagnosis that precludes participation
* dementia
* under the care of another multi-disciplinary clinic.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — self identified as women
Enrollment: 50 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
health self efficacy | 6 months after intervention initiation
  self report measure adapted from Moore and McBride 2009 that consists of 2 questions, on a scale of 0-10, how much do i want change and how much am I capable of change, with 10 reflecting higher self efficacy
goal adherence | average of monthly measures at months 1-6.
  Goal Attainment Scale for rehabilitation. This is scaled from -3 to +2, with +2 representing goal attainment far beyond anticipated, 0 representing goal achievement and -2 representing worsening. Higher is better.

SECONDARY OUTCOMES:
weight | 6 months after intervention inititiation
  kg
cardiovascular risk | 6 months after intervention initiation
  hebrew adapted Healthy Heart Score which includes assessment of physical activity, nutrition behaviors, smoking and alcohol consumption
experiential avoidance | 6 months after intervention initiation
  Brief Experiential Avoidance Questionnaire This is a 15 item scale with answers that range from 1-6 with scores ranging from 15-90 with higher scores reflecting more avoidance
blood pressure | 6 months after intervention initiation
  systolic and diastolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Donna R Zwas, MD MPH, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Yes
Partially, with masking of psychological information, only to researchers with GCP upon request.
Supporting Information: Study Protocol, ICF
Time Frame: upon publication
Access Criteria: GCP, upon request